CLINICAL TRIAL: NCT02167815
Title: A Multicenter, Post Marketing Clinical Follow up (PMCF) Investigation to Evaluate the Performance and Safety of a Soft Silicone Foam Dressing and to Evaluate the Performance of Standard Care in Exuding Venous Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RedEgg 01
Record Dates: First submitted 2014-05-15; First posted 2014-06-19 (Estimated); Results first posted 2016-10-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2014-05

CONDITIONS: Venous Leg Ulcer (VLU)
MeSH Terms: conditions — Varicose Ulcer | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (Active Comparator): standard care ( such as alginate, hydrofiber or other treatment)
  Interventions: Other: standard care
- Intervention ( Mepilex XT) (Experimental)
  Interventions: Device: Mepilex XT

INTERVENTIONS:
Device: Mepilex XT — Experimental arm
  Arms: Intervention ( Mepilex XT)
Other: standard care
  Arms: Standard care

SUMMARY:
This investigation is a Post Marketing Follow-Up Study for Mepilex XT conducted as part of Mölnlycke Health Care's quality system. The primary objective is to evaluate the performance of the dressing when used as intended on exuding Venous Leg Ulcers (VLUs) in the inflammatory and granulating stages of the wound healing process.

ELIGIBILITY:
Inclusion Criteria:

1. Venous Leg Ulcer
2. Exuding wound
3. Wound surface covered with sloughy tissue* (before debridement)
4. Wound size ≥ 6 cm2
5. In case of multiple wounds, target wound must be ≥ 3cm distant from other wounds.
6. Wound suitable for treatment with the relevant primary dressing**
7. Male or female, 18 years of age and above
8. Signed Informed Consent

   * Sloughy tissue defined as wet, yellow-brown fibrinous tissue present in the wound bed ** Mepilex XT in the intervention group. Standard care in the observation group

Exclusion Criteria:

1. More than two products of 15 cm x15 cm needed to cover the whole wound and affected peri-wound area
2. Wound cavity and/or fistula
3. Full thickness burns
4. Exposed tendons and/or fascia
5. Bleeding wounds
6. Malignant or fungating wounds
7. Wound age > 12 months
8. Use of antimicrobial dressings or topical agents such as antiseptics, local antibiotics and steroids within 7 days from inclusion on the wound intended to be included
9. Untreated limb ischemia (according to investigator's judgement) at the time of inclusion
10. Subject not suitable for the investigation according to the investigator's judgement
11. Subject included in other ongoing clinical investigation which could interfere with this investigation, as judged by the investigator
12. Known allergy/hypersensitivity to any of the components of the primary dressing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Czechia (3):
  - Nemocnice Podlesí a.s., Třinec, Konská 453
  - Nemocnice Jihlava, Jihlava, Vrchlického
  - The General University Hospital in Prague, Prague

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Care: standard care ( such as alginate, hydrofiber or other treatment)
  standard care
Period: Overall Study
Arm/Group | Standard Care | Intervention ( Mepilex XT)
Started | 9 | 21
Completed | 9 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that have used at least one product and that have some follow-up data for the primary endpoint is included in the population presented.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Intervention ( Mepilex XT) | Total
Number analyzed (Participants) | 9 | 21 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 10 | 15
  >=65 years | 4 | 11 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 4 | 12 | 16
Region of Enrollment [Number; unit: participants]
  Czech Republic | 9 | 21 | 30

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline in Condition of the Peri Wound Skin
Description: Deteriorationin of skin condition , Mepilex XT and Standard care (%)
Time Frame: 16 weeks
Population: Intention to treat, change from baseline in condition of the peri-wound skin.
Measure: Number; unit: percentage of subjects
Groups:
- Standard Care: observation group, treating according to investigation sites standard care
Arm/Group | Intervention ( Mepilex XT) | Standard Care
Number analyzed (Participants) | 21 | 9
percentage of subjects
  Redness | 0 | 0
  Rash | 5.6 | 16.7
  Maceration | 11.1 | 16.7
  Dermatitis | 0 | 16.7
  Blistering | 0 | 0
  skinstripping | 5.6 | 0
  Trauma to wound edges | 5.6 | 0
  Product degradation | 16.7 | 16.7

2. Secondary Outcome: Pain Scores on the Visual Analog Scale
Description: Pain at baseline visit, compared with pain at week 16. VAS scale, minimum pain = 0, maximum pain = 100.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale (VAS)
Groups:
- Standard Care: observation group, treated according to investigation sites standard care
Arm/Group | Intervention ( Mepilex XT) | Standard Care
Number analyzed (Participants) | 21 | 9
units on a scale (VAS)
  Pain at baseline | 17.6 (12.6) | 24.0 (22.2)
  Pain at week 16 | 5.8 (14.2) | 12.0 (21.7)

3. Secondary Outcome: Users Feedback After Handling or Use as a Measure of Performance.
Description: Investigator/Nurse and Subject evaluation of performance of the primary dressing ( n) Scale= Good , Very Good, Poor, Very Poor
  1Ease of application, 2 Ease of removal, 3 Ability to retain exudate, 4 Adherence to healthy skin, 5 Confomability to be repositioned , 6 Overall satisfaction, 7 Dressing sticking to wound bed, 8 Presence of residues on the wound bed. 9 Presence of residues on the healthy skin. 10 Overall evaluation of change in periwound skin condition.
Time Frame: 16 weeks
Measure: Number; unit: participants
Groups:
- Standard Care: observation group, treated according to investigation sites, standard care
Arm/Group | Intervention ( Mepilex XT) | Standard Care
Number analyzed (Participants) | 21 | 9
participants
  Baseline Ease of application good/very good | 21 | 9
  Baseline Ease of removal good/very good | 5 | 6
  Baseline Ease of removal poor/very poor | 0 | 3
  Baseline Ability to retain exudate good/very good | 21 | 4
  Baseline Ability to retain exudate poor | 0 | 5
  Baseline Adherence to healthy skin good/very good | 21 | 5
  Baseline Adherence to healthy skin poor/very poor | 0 | 4
  Baseline conformability good/very good | 21 | 8
  Baseline conformability poor | 0 | 1
  Baseline ability to be reposition good/very good | 19 | 8
  Baseline ability to be reposition very poor/poor | 1 | 1
  Baseline overall satisfaction good/very good | 21 | 8
  Baseline overall satisfaction poor/very poor | 0 | 1
  Baseline sticking to woundbed moderate/high | 0 | 5
  Baseline sticking to woundbed none/low | 21 | 4
  Baseline pressens of residues wound moderate | 0 | 1
  Baseline pressens of residues wound none/low | 21 | 7
  Baseline pressens of residues skin none/low | 21 | 9
  Last visit, ease of removal good/very good | 18 | 4
  Last visit, ease of removal poor | 0 | 1
  Last visit, retain exudate good/very good | 17 | 1
  Last visit, retain of exudate poor | 0 | 4
  Last visit, adherence to skin good/very good | 17 | 4
  Last Visit, adherence to skin poor | 1 | 1
  Last Visit, conformability good/very good | 18 | 4
  Last visit, conformability poor | 0 | 1
  Last Visit, ability to be reposition good/very goo | 18 | 4
  Last Visit, ability to be reposition poor | 0 | 1
  Last visit, overal satisfaction good/very good | 18 | 4
  Last visit, overal satisfaction poor | 0 | 1
  Last visit, sticking to the wound moderate/low | 4 | 5
  Last visit, sticking to the wound none | 14 | 0
  Last visit, presence of residues wound none/low | 18 | 5
  Last visit, presence of residues skin none | 18 | 4
  Last visit, presence of residues skin moderate | 0 | 1
  Last visit, change in periwound condition improved | 14 | 5
  Last visit, change in periwound skin unchanged | 3 | 1
  Last visit, change in periwound skin, deteriorated | 1 | 0

4. Secondary Outcome: Measure of Actual Dressing Cost and Cost of Care, as Input for Health Economics Calculations.
Time Frame: 16 weeks
Population: the way to collect data differed to much betwen the sites, no analysis could be done.
Arm/Group | Intervention ( Mepilex XT)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Standard Care | Intervention ( Mepilex XT)
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/21
Other Adverse Events (participants affected / at risk) | 0/9 | 3/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=9) | Intervention ( Mepilex XT) (N=21)
Low pain in the skin under dressing (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) — unlikely relattionship to dressing
wound infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — superficial wound infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less